CLINICAL TRIAL: NCT06335212
Title: Peripheral Defocus Profile of Multifocal Minus Contact Lenses
Status: Completed | Type: Observational
Sponsor: State University of New York College of Optometry (Other)
Responsible Party: Principal Investigator, Xiaoying Zhu, OD, PhD, MD, MS, FAAO, Assistant Clinical Professor, State University of New York College of Optometry
Other Study IDs: IRBNET ID 1448963
Record Dates: First submitted 2022-12-26; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Myopia; Refractive Errors; Contact Lens
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- One group of subjects were recruited.
  Interventions: Device: Single vision and multifocal contact lenses

INTERVENTIONS:
Device: Single vision and multifocal contact lenses — Cycloplegic central autorefraction was conducted with both Grand Seiko WAM-5500 open-field auto-refractor (Grand Seiko Co Ltd) and OPD OPD-Scan III Wavefront Aberrometer (Marco) on the subjects in the following conditions: (1) no CLs, (2) SVCLs, (3) MFCLs (+2.00D Add), and (4) MFCLs (+4.00D Add). Relative peripheral power profiles were measured using the OPD under the same 4 conditions after cycloplegia.

SUMMARY:
Purpose: Numerous studies have proven that emmetropization in young animals including humans is regulated by visual input. It has long been hypothesized that peripheral myopic defocus may act as a stop signal to reduce myopia progression and axial elongation. As such, multifocal soft contact lenses (MFCLs) have been utilized for myopia control in school-aged children, with variable efficacies. One potential explanation is that the actual peripheral myopic defocus an eye experiences during MFCL wear may not be identical to the Add power and not sufficient to reduce myopia progression. Our study investigated and compared the peripheral power profiles of myopic eyes when they were uncorrected and wore single vision contact lenses (SVCLs) and MFCLs of different Add powers.

Methods: Subjects with -1.00 D to -10.00 D of myopia (SE, determined with manifest refraction) were custom fit with both single vision (SV) and MFCLs (+2.00 and +4.00 D Add; provided by Specialeyes) in both eyes. These Specialeyes MFCLs had an aspheric design with a standard total optical zone of 8.0mm. Cycloplegic central autorefraction was conducted with both Grand Seiko WAM-5500 open-field auto-refractor (Grand Seiko Co Ltd) and OPD OPD-Scan III Wavefront Aberrometer (Marco) on the subjects in the following conditions: (1) no CLs, (2) SVCLs, (3) MFCLs (+2.00D Add), and (4) MFCLs (+4.00D Add). Relative peripheral power profiles were measured using the OPD under the same 4 conditions after cycloplegia. Data in the right eye was used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* spherical equivalent (determined with subjective refraction) between -1.00 and -10.00 D in each eye, spherical power between -0.75 and -10.00 D and cylindrical power ≤ 1.50 D
* monocular best corrected visual acuity 20/25 or better
* no previous contact lens experience required
* no history of ocular pathology, binocular vision anomalies, or refractive surgery.

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults between 18 and 30 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
refractive power | Relative pupil limited optical power profile was measured once within one month from their first visit when the subjects were uncorrected or wearing contact lenses of various designs
  Relative pupil limited optical power profile

CONTACTS AND LOCATIONS:
Locations (1):
- State University of New York, College of Optometry, New York, New York, United States